CLINICAL TRIAL: NCT06848790
Title: Effectiveness of Different Methods of Interdental Space Hygiene in Daily Practice Among Young Adults: A Randomized, Single-Blind Controlled Trial
Brief Title: Interdental Hygiene Methods in Young Adults
Acronym: HIJA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 69HCL24_1272
Record Dates: First submitted 2025-02-17; First posted 2025-02-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Microbiota-related Disease; Oral Hygiene; Periodontal Diseases
Keywords: Oral health; Interdental hygiene; Periodontal disease prevention; Interdental microbiota; Preventive care
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calibrated interdental brush (Experimental): Healthy adult volunteers (not suffering from chronic pathologies) and non-smokers, agreeing to change their interdental hygiene habits for 3 months by daily using a calibrated interdental brushes .
  Interventions: Procedure: Calibrated interdental brush
- Non-calibrated interdental brush (No Intervention): Healthy adult volunteers (not suffering from chronic pathologies) and non-smokers, agreeing to change their interdental hygiene habits for 3 months by daily using a non-calibrated interdental brushes .

INTERVENTIONS:
Procedure: Calibrated interdental brush — participants will use calibrated interdental brushes
  Arms: Calibrated interdental brush

SUMMARY:
Oral health is essential for overall well-being and systemic health. A key factor in preserving this health is maintaining the balance of the interdental microbiota, which involves regulating the quantity of pathogenic bacteria in interdental spaces (IS). These IS represent a unique ecological niche where the body has limited specific defense mechanisms, making them vulnerable to infections.

In adults, the colonization of interdental spaces by pathogenic bacteria increases the risk of periodontal diseases, which are themselves associated with non-communicable diseases such as cardiovascular diseases, diabetes, and certain types of cancer.

Preventing interdental microbiota dysbiosis from a young age is therefore a priority to maintain quality oral health and contribute to good systemic health throughout life. However, conventional brushing techniques cover only accessible tooth surfaces and cannot reach the interdental spaces. Currently, the use of interdental brushes (IDBs) is recognized as the most effective method for interdental hygiene. There are various types of IDBs, differing in several aspects that influence their effectiveness and usability. The main differences relate to their shape, size, and calibration using an interdental probe or not, allowing adaptation to different interdental space sizes. To date, only one study has demonstrated the effectiveness of daily calibrated interdental brush use in reducing dysbiosis and interdental inflammation among young adults. However, no research has yet been conducted to compare the effectiveness of the various types of IDBs available on the market (calibrated versus non-calibrated).

ELIGIBILITY:
Inclusion Criteria:

* Person between 18 and 30 years old
* Person who has given free, informed, express written consent
* Person affiliated to a French social security system
* Person living or working in Lyon or the Lyon conurbation served by public transport (TCL)

Exclusion Criteria:

* Person with a smoking addiction
* Person participating in another study related to oral hygiene
* Patients at high risk of infective endocarditis
* Person with chronic pathologies
* Person having taken antibiotic treatment during the month preceding the start of the study
* Pregnant, parturient or breastfeeding woman
* Persons deprived of liberty by a judicial or administrative decision
* People receiving psychiatric care
* Persons admitted to a health or social establishment for purposes other than research
* Adults subject to a legal protection measure (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
* Person with fewer than 20 natural teeth
* Person performing interdental hygiene and/or daily mouthwashes.
* Person wearing orthodontic appliance
* Person with periodontal disease (stage ≥ II periodontal lesions according to the Chicago 2017 classification (i.e. PD ≥ 4 mm, and/or CAL ≥ 4 mm) and/or generalized (>30% of sites )), active caries or during dental care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-06-17 (Estimated)

PRIMARY OUTCOMES:
Interdental bleeding at month 3 (in percentage) | Baseline (T0), 3 months after baseline (T3)
  Comparison of interdental inflammation (interdental bleeding) following the daily use of calibrated versus non-calibrated interdental brushes at month 3 (T3, expressed as a percentage and assessed at four sites per tooth following probing with a periodontal probe).

SECONDARY OUTCOMES:
Composition of the Interdental microbiome (diversity and total bacteria count) | Baseline (T0)
  Identification of the composition of the interdental microbiome in healthy young adults using sequencing techniques at T0, in four standardized sites (between teeth 15-16, 25-26, 35-36, and 45-46). If the specified teeth are missing, exhibit pathologies, or have diastemas preventing interdental cleaning, the sample will be taken from the nearest healthy mesial interdental space.
Periodontal health analysis | Baseline (T0), 1 week later (T1), 1 month after baseline (T2), 3 months after baseline (T3)
  Comparison of periodontal for all participant's teeth (plaque index, gingival index, interdental inflammation, pocket depth and loss of clinical attachment) before (T0), 1 week after baseline (T1), 1 month after baseline (T2) and 3 months after baseline (T3) following the daily use of calibrated versus non-calibrated interdental brushes
Periodontal health analysis - salivary pH | Baseline (T0), 1 week later (T1), 1 month after baseline (T2), 3 months after baseline (T3)
  Comparison of periodontal for all participant's teeth (salivary pH) before (T0), 1 week after baseline (T1), 1 month after baseline (T2) and 3 months after baseline (T3) following the daily use of calibrated versus non-calibrated interdental brushes
Interdental microbiota at T3 (diversity and total bacteria count) | Baseline (T0), 3 months after baseline (T3)
  Comparison of the composition of the interdental microbiome in healthy young adults using sequencing techniques after 3 months of calibrated versus non calibrated interdental brushed, in four standardized sites (between teeth 15-16, 25-26, 35-36, and 45-46). If the specified teeth are missing, exhibit pathologies, or have diastemas preventing interdental cleaning, the sample will be taken from the nearest healthy mesial interdental space.
Daily use acceptability of interdental brushes | 1 week after baseline (T1), 1 month after baseline (T2), 3 months after baseline (T3)
  Evaluation and comparison of the acceptability and ease of integration (by TFA questionnaire) of daily use of calibrated versus non-calibrated interdental brushes, 1 week after baseline (T1), 1 month after baseline (T2) and 3 months after baseline (T3)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane VIENNOT, Principal Investigator — HCL
Locations (1):
- Service de Soins Dentaires Et D'Odontologie, Lyon, France